CLINICAL TRIAL: NCT02807818
Title: The Effects on Early Brain Development of a Nurse Home Visitation Program for Pregnant Youth and Their Families Living in a Poor Urban Area in Sao Paulo, Brazil
Brief Title: A Home Visiting Program for Pregnant Youth to Promote Early Brain Development
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Guilherme Vanoni Polanczyk, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0722-03
Record Dates: First submitted 2016-06-09; First posted 2016-06-21 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Child Development
Keywords: Child development; Infant; Mother-Child Relations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nurse home visits (Experimental): Nurse biweekly home visit.
  Interventions: Behavioral: Home visiting Program for Young Pregnant Women
- Usual care (No Intervention): Usual care.

INTERVENTIONS:
Behavioral: Home visiting Program for Young Pregnant Women
  Arms: Nurse home visits

SUMMARY:
Home visiting programs for pregnant women aiming to improve mother-infant relationship has received worldwide attention in the past 30 years. These programs are considered an important strategy to improve women's health during pregnancy, aside from improving child's birthing conditions and allowing parents access to tools which will nurture and properly stimulate their baby, thus promoting emotional and cognitive development. Objectives: The "Nurse home visitation program for pregnant youth" aims to promote infant´s healthy development, from pregnancy to the first months of life, in a high-risk population. Methods: Eighty young pregnant women aged between 14 and 20 years were randomly allocated to the intervention or to usual prenatal care program. The "Nurse home visitation program for pregnant youth" was developed based on Albert Bandura's theory of self-efficacy, on Urie Bronfenbrenner´s bioecological model, which recognizes the importance of individual and family inclusion in various contexts of social life, on John Bowlby and Mary Ainsworth evolutionary theories of attachment, which involves the care practitioner addressing issues such as environmental health, life course and parenting, bond between mother and infant, and infant´s social and cognitive development. Neuropsychomotor development will be assessed at 3, 6 and 12 months using the Bayley Scale of Infant Development. Brain development will be assessed via electroencephalography at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Low socioeconomic status
* Mother's age between 14-19
* Mother being a primapara
* Gestation between the 8th and 16th week

Exclusion Criteria:

* High-risk gestation
* Mother's Intellectual, visual or auditory disability

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in neuropsychomotor development during first year of life | From 3 to 12 months of age
  Complete child assessment with the Bayley Scale of Infant Development at 3, 6 and 12 months of age.

SECONDARY OUTCOMES:
Change in child brain maturation | At 6 and 12 months
  Assessment of brain wave patterns (alpha, gamma and theta frequencies) via electroencephalography (EEG).
Mother-child attachment biomarker | At 6 and 12 months
  Assessment of event-related potential associated with child face recognition of the mother via electroencephalography (EEG).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] da Silva LA, Siqueira LD, Oliveira LGF, Miguel Filho EC, Polanczyk GV, Fracolli LA. The impact of a home visiting program on the care environment of Brazilian adolescent mothers - an descriptive exploratory study. Front Glob Womens Health. 2025 Apr 25;6:1530351. doi: 10.3389/fgwh.2025.1530351. eCollection 2025. PMID 40351759
- [Derived] Euclydes VLV, Gastaldi VD, Feltrin AS, Hoffman DJ, Gouveia G, Cogo H, Felipe-Silva A, Vieira RP, Miguel EC, Polanczyk GV, Chiesa A, Fracolli L, Matijasevich A, Ferraro A, Argeu A, Maschietto M, Brentani HP. DNA methylation mediates a randomized controlled trial home-visiting intervention during pregnancy and the Bayley infant's cognitive scores at 12 months of age. J Dev Orig Health Dis. 2022 Oct;13(5):556-565. doi: 10.1017/S2040174421000738. Epub 2022 Mar 8. PMID 35256034
- [Derived] Fatori D, Fonseca Zuccolo P, Shephard E, Brentani H, Matijasevich A, Archanjo Ferraro A, Aparecida Fracolli L, Chiesa AM, Leckman J, Constantino Miguel E, V Polanczyk G. A randomized controlled trial testing the efficacy of a Nurse Home Visiting Program for Pregnant Adolescents. Sci Rep. 2021 Jul 13;11(1):14432. doi: 10.1038/s41598-021-93938-7. PMID 34257407
- [Derived] Alarcao FSP, Shephard E, Fatori D, Amavel R, Chiesa A, Fracolli L, Matijasevich A, Brentani H, Nelson CA, Leckman J, Miguel EC, Polanczyk GV. Promoting mother-infant relationships and underlying neural correlates: Results from a randomized controlled trial of a home-visiting program for adolescent mothers in Brazil. Dev Sci. 2021 Nov;24(6):e13113. doi: 10.1111/desc.13113. Epub 2021 Apr 12. PMID 33844435
- [Derived] Fatori D, Argeu A, Brentani H, Chiesa A, Fracolli L, Matijasevich A, Miguel EC, Polanczyk G. Maternal Parenting Electronic Diary in the Context of a Home Visit Intervention for Adolescent Mothers in an Urban Deprived Area of Sao Paulo, Brazil: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Jul 28;8(7):e13686. doi: 10.2196/13686. PMID 32720906